CLINICAL TRIAL: NCT01267968
Title: An Open-label, Randomized, Single Period, Parallel-Cohort Study To Evaluate Serum and Pulmonary Pharmacokinetics Following Single and Multiple Dose Administration of Intravenous GSK2251052 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 114926
Record Dates: First submitted 2010-12-16; First posted 2010-12-29 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Community-acquired Infection
Keywords: pharmacokinetics; bronchoalveolar lavage; GSK2251052; pulmonary; healthy volunteer; antimicrobial
MeSH Terms: conditions — Community-Acquired Infections | interventions — 3-(aminomethyl)-7-(3-hydroxypropoxy)-1-hydroxy-1,3-dihydro-2,1-benzoxaborole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): GSK2251052 1500 mg Single dose (i.v., 60 min)
  Interventions: Drug: GSK2251052
- Cohort 2 (Experimental): GSK2251052 1500 mg IV q12h x 5 doses infused over 60 minutes
  Interventions: Drug: GSK2251052

INTERVENTIONS:
Drug: GSK2251052 — 1500 mg (dosing detailed in Arm description)

SUMMARY:
GSK2251052 is a member of a novel mechanistic and structural class of antibiotics that inhibits the bacterial enzyme leucyl tRNA synthetase (LeuRS) by forming a boron adduct with tRNA and is currently in development for the treatment of hospital acquired Gram-negative infections (including E. coli, K. pneumoniae, and Enterobacter spp.).

This is an open-label, randomized, single period, parallel-cohort pharmacokinetic study to evaluate serum and pulmonary pharmacokinetics following single dose and multiple dose administration of intravenous GSK2251052. In Cohort 1, approximately 15 healthy adult subjects will be randomized to receive a single IV dose of GSK2251052 1500 mg in the fasted state. Following the dose, bronchoalveolar lavage (BAL) fluid and serial plasma samples will be collected for determination of GSK2251052 parent and metabolite concentrations. In Cohort 2, approximately 15 healthy adult subjects will receive GSK2251052 1500 mg IV BID x 5 doses (Cohort 2). Following the last dose in the fasted state, bronchoalveolar lavage (BAL) fluid and serial plasma samples will be collected for determination of GSK2251052 parent and metabolite concentrations. Vital signs, ECGs, and adverse events will be monitored throughout the study. A follow up visit will occur 10 to 14 days after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphatase and bilirubin < or = 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). Abnormal LFT tests may be repeated once at the discretion of the Investigator. If an abnormality is repeated, the subject would not be eligible for inclusion.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and ECGs. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea. A follicle stimulating hormone (FSH) will be performed for confirmation. For this study, FSH level > 40 MlU/ml is confirmatory].
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until the follow-up visit.
* Body weight > or = 50 kg for men and > or = 45 kg for women and BMI within the range 18.5-30.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* QTcB or QTcF <450 msec or QTcB or QTcF <480 msec in subjects with Bundle Branch Block.

Exclusion Criteria:

* Deviations from exclusion criteria are not allowed because they can potentially jeopardize the scientific integrity of the study, regulatory acceptability or subject safety. Therefore, adherence to the criteria as specified in the protocol is essential.
* A subject will not be eligible for inclusion in this study if any of the following criteria apply:
* Contraindications to bronchoalveolar lavage including hypercapnia >50 mm Hg, refractory hypoxemia, reactive airway disease or asthma, unstable angina or acute myocardial infarction in the last 6 months, heart failure, and severe hemostatic alterations.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids, and benzodiazepines.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* History of sensitivity to pre- and post-procedure medications related to the BAL procedure such as codeine, atropine, lidocaine, midazolam, and fentanyl.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive urine hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice [and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices] from 7 days prior to the first dose of study medication.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination): Heart rate < 45 and > 100 bpm (males), < 50 and > 100 bpm (females); PR interval <120 and > 220 msec; QTcB interval >450 msec
* Evidence of previous myocardial infarction (does not include ST segment changes associated with repolarization).
* Any conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree or higher], Wolf Parkinson White [WPW] syndrome), sinus pauses> 3 seconds, non-sustained or sustained ventricular tachycardia (≥3 consecutive ventricular ectopic beats) or any significant arrhythmia which, in the opinion of the principal investigator and GSK medical monitor, will interfere with the safety of the individual subject.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2011-01-11 (Actual); Primary Completion 2011-03-16 (Actual); Study Completion 2011-03-16 (Actual)

PRIMARY OUTCOMES:
Epithelial lining fluid (ELF)/ plasma ratios for GSK2251052 at early, mid, and late dosing interval timepoints following intravenous administration of 1500 mg q12h. | up to 3 days
Alveolar macrophage (AM)/ plasma ratios for GSK2251052 at early, mid, and late dosing interval timepoints following intravenous administration of 1500 mg q12h. | up to 3 days

SECONDARY OUTCOMES:
Plasma AUC (0-t), Cmax, CL, Vss, and t½, following intravenous administration of GSK2251052, as permitted by the data. | up to 3 days
GSK2251052 concentrations in urine following single and repeat dose administration | up to 3 days
Safety and tolerability parameters, including adverse event, concurrent medication, clinical laboratory, cardiac monitoring, and vital signs assessments. | up to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Tenero D, Bowers G, Rodvold KA, Patel A, Kurtinecz M, Dumont E, Tomayko J, Patel P. Intrapulmonary pharmacokinetics of GSK2251052 in healthy volunteers. Antimicrob Agents Chemother. 2013 Jul;57(7):3334-9. doi: 10.1128/AAC.02483-12. Epub 2013 May 6. PMID 23650164
- See also: Results for study 114926 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114926?search=study&search_terms=114926#rs